CLINICAL TRIAL: NCT00608192
Title: HIV and Hepatitis Care Coordination in Methadone Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: R01DA020781 (NIH); R01DA020781 (NIH)
Record Dates: First submitted 2008-01-18; First posted 2008-02-06 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Hepatitis, Viral, Human; HIV Infections
Keywords: HIV; viral hepatitis; methadone maintenance; case management; costs; vaccination; risk reduction education
MeSH Terms: conditions — Hepatitis, Viral, Human; HIV Infections | interventions — Educational Status; Counseling

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Testing, Education, & Counseling (TEC) (Active Comparator): HIV and hepatitis screening is done on-site, but vaccination and medical care will be provided by off-site referral. HIV and Hepatitis, Testing, Education, & Counseling (TEC) participants will receive standard HIV and hepatitis education & counseling. TEC participants will not receive case management services.
  Interventions: Behavioral: Testing, Education, & Counseling (TEC)
- Hepatitis Care Coordination (HCC) (Experimental): Participants will receive on-site HIV and viral hepatitis screening. Hepatitis A and B combination vaccination will be provided on-site. Participants will receive on-site theory-based HIV and hepatitis education, counseling, and 6 months of case management to promote adherence to HIV and HCV evaluation.
  Interventions: Behavioral: Hepatitis Care Coordination (HCC)

INTERVENTIONS:
Behavioral: Testing, Education, & Counseling (TEC) — Trained research staff will provide a two-session HIV/hepatitis education class. Participants will also be offered serological testing for hepatitis A, B and C, and HIV (optional), and off-site referrals for vaccination and hepatitis care. The content of the TEC intervention is evidence based. The TEC condition is comparable to screening and education methods commonly used in many drug treatment settings. Those in the TEC intervention group who do not adhere to needed off site vaccinations will be offered on site vaccination 30 days after vaccination referral.
  Arms: Testing, Education, & Counseling (TEC)
Behavioral: Hepatitis Care Coordination (HCC) — HCC Participants will be offered serological testing and counseling for hepatitis A, B and C, and HIV (optional). HCC participants will be offered on-site hepatitis A and B combination vaccination at the methadone clinic. They will also receive a two-session HIV/hepatitis education class with Motivational Interviewing. In addition, participants will receive 6 months of weekly case management to facilitate entry into hepatitis care.
  Arms: Hepatitis Care Coordination (HCC)

SUMMARY:
This randomized clinical trial will examine the effectiveness of a strategy of HIV and Hepatitis Care Coordination (HCC) consisting of testing, education, counseling and vaccination for methadone maintenance patients compared with standard Testing, Education, and Counseling (TEC).

DETAILED DESCRIPTION:
In the HCC model, HIV and hepatitis screening, and HAV and HBV vaccination will be done on site and participants receive on site theory-based HIV and hepatitis education, counseling, and case management to promote adherence to HIV and HCV evaluation; in TEC hepatitis screening is done on site, but vaccination and medical care will be provided by off site referral. Primary aims are to assess the impact of the HCC intervention on adherence to hepatitis A virus (HAV) and hepatitis B virus (HBV) vaccination and attendance at an initial appointment with an HIV and/or HCV care provider. Secondary aims include examining intervention effects on HIV and hepatitis knowledge, risky behaviors, alcohol use; follow-up with later stages of HIV and hepatitis C care; to identify psychological mediators of intervention outcomes; and to estimate the incremental cost of the HCC intervention to facilitate fuller economic evaluations of the intervention if proven effective.

ELIGIBILITY:
Inclusion Criteria:

* >=18 years of age
* be able to provide informed consent
* agree to participate in hepatitis/HIV intervention
* expect to be available to participate in the study for the entire duration of the study
* HCV negative, of unknown HCV status, or have not received any previous medical care for HCV

Exclusion Criteria:

* have already had a formal hepatitis C evaluation
* are obtaining medical care for hepatitis C
* not interested in obtaining medical care for hepatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 489 (Actual)
Dates: Start 2008-01; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Vaccination adherence visits | 30 days
Health Care Utilization Survey | 12 months
Intervention Costs & Hepatitis Care Utilization: DATCAP, public and private health care system administrative databases | 12 months

SECONDARY OUTCOMES:
Hepatitis A Knowledge Test | post-intervention & 90 days
Hepatitis B Knowledge Test | post-intervention & 90 days
Hepatitis C Knowledge Test | post-intervention & 90 days
HIV Knowledge Test | post-intervention & 90 days
Risk Behavior Survey | 3 months, 9 months, 12 months
Addiction Severity Index | 3 months, 9 months, 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Carmen L Masson, Ph.D., Principal Investigator — Univerisity of California, San Francisco, Dept. of Psychiatry; David Perlman, MD, Principal Investigator — Chemical Dependency Institute at Beth Israel Medical Center
Locations (2):
- United States (2):
  - San Francisco General Hospital Opiate Treatment Outpatient Program, San Francisco, California
  - Beth Israel Medical Center Methadone Maintenance Program, New York, New York